CLINICAL TRIAL: NCT06195332
Title: Comparison of Open and Endoscopic Transversus Abdominis Release for Midline Incisional Ventral Hernia - a Randomized Controlled Trial
Brief Title: Open Vs. Endoscopic Transversus Abdominis Release Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City Clinical Hospital No.1 named after N.I. Pirogov (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2907-2/22
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Incisional Hernia of Midline of Abdomen
Keywords: incisional hernia; eTEP; open TAR; endoscopic TAR; transversus abdominis release
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- open TAR (Active Comparator): Open transversus abdominis release procedure will be use as combine open procedure Rives-Stoppa hernia repair in combination with bilateral transversus abdominis release with retromuscular mesh placement
  Interventions: Procedure: open TAR
- endoscopic TAR (Active Comparator): Endoscopic transversus abdominis release procedure will be use as combine minimally invasive Rives-Stoppa hernia repair in combination with bilateral transversus abdominis release via endoscopic technique with retromuscular mesh placement
  Interventions: Procedure: endoscopic TAR

INTERVENTIONS:
Procedure: open TAR — Participants will undergo open TAR repair according to the assigned treatment arm.
  Other Names: open transversus abdominis release
  Arms: open TAR
Procedure: endoscopic TAR — Participants will undergo endoscopic TAR repair according to the assigned treatment arm.
  Other Names: endoscopic transversus abdominis release
  Arms: endoscopic TAR

SUMMARY:
This study aims to comparatively evaluate the early and long-term results of open and endoscopic TAR procedure for large midline incisional ventral hernias.

DETAILED DESCRIPTION:
Minimally invasive (endoscopic) transversus abdominis release (TAR) - new technique for the treatment of patients with large incisional ventral hernia. Term "endoscopic" TAR combines two minimally invasive (laparosopic or extraperitoneal (eTEP) approaches. These techniques have demonstrated significant advantages compared with open TAR in several retrospective studies. There are currently no randomized trials comparing open and endoscopic TAR operations for incisional ventral hernia repair.This study aims to comparatively evaluate the early and long-term results of open and endoscopic TAR procedure for large midline incisional ventral hernias.

The sample size was determined based on a previously conducted retrospective pilot study comparing the results of open and endoscopic TAR procedures for midline incisional ventral hernia repair. The retrospective study included 133 patients with midline incisional ventral hernias who were underwent Rives-Stoppa hernia repair in combination with bilateral posterior component separation with transversus abdominis release via open (open TAR) or endoscopic (eTAR) technique in Moscow City Hospital №1 from January 2018 to December 2022. All patients were included in the study, starting from the moment of endoscopic TAR technique was introduced into the clinic. At the same time, the learning curve for the open TAR had already been reached at that time; more than 20 open TAR interventions were performed in the clinic in 2016-2017. The average hospitalization time in open TAR group was 6.7 ± 2.14 days. In endoscopic TAR group the average hospitalization time after surgery was 5.2 ± 1.65 bed days. After achieving the learning curve (20 operations) for the endoscopic TAR procedure technique average hospitalization period after surgery was 4.8 ± 1.47 days. Thus, a decrease in the duration of hospitalization in endoscopic TAR group after reaching the learning curve was noted by 28.4%. This fact, based on a retrospective pilot study, allows the investigators to assume as a hypothesis for this RCT a reduction in the duration of hospitalization during endoscopic TAR by at least 30% as a guideline for calculating the power of the study. Thus, assuming a Type I error probability α of 0.05 and a Type 2 error probability β of 0.20, it would require a total sample size of 36 patients (18 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

* midline incisional hernia
* defect width from 8 till 12 cm
* ASA I-III class
* able to give informed consent
* elective hernia repair
* considered eligible for minimally invasive ventral hernia repair

Exclusion Criteria:

* primary ventral hernia
* lateral hernia with/without midline
* refuse to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
length of stay after surgery | 30 days after surgery
  From date of operation until discharge

SECONDARY OUTCOMES:
duration of operation | period of operation
  time from beginning to the end of surgery
surgical site occurrences rate | 30 days after surgery
  incidence of all type of wound complications
surgical site infection rate | 30 days after surgery
  incidence of wound infection
rate of postoperative complications | 30 days after surgery
  number of participants with postoperative complications
rate of postoperative complications Clavien 3a and higher | 30 days after surgery
  number of participants with postoperative complications Clavien 3a and higher, evaluated by Clavien-Dindo classification of surgical complications from Dindo et al.
Comprehensive complication index | 30 days after surgery
  Comprehensive complication index will be calculated after verification of all complications and their classification according to Clavien, evaluated by Clavien-Dindo classification of surgical complications from Dindo et al. Minimum (0 points) - best results, maximum (100 points) - worst result (patient death)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical City Hospital #1 named after N.I. Pirogov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No